# Low-Dose Atropine for Treatment of Myopia (Myopia Treatment Study)

Informed Consent Form April 16, 2019

NCT03334253



# CONSENT FOR YOUR CHILD TO TAKE PART IN A RESEARCH STUDY

**STUDY TITLE:** Low-Dose Atropine for Treatment of Myopia (MTS1)

| 010212001011011011 |
|---------------------------------|
| Name: |
| Contact Number: |
| Site Name: |
| Site Address: |
| Emergency (24-hour) Number: |
| Study Coordinator Name/Contact: |

STUDY DOCTOR'S INFORMATION

#### **SUMMARY**

This consent form will give you important information about this study. It will help you decide if would like to allow your child to take part in the study. You do not have to allow your child to be in this study. You or your child can decide to stop being in the study at any time. You should read and discuss all the information in this consent form with the study doctor and your child.

- The study is being done to see if low-dose eye drops of a drug called atropine can help prevent myopia (nearsightedness) from getting worse. Atropine is not approved by the FDA for treating myopia. It is considered an experimental drug when being used to treat myopia.
- We are asking that your child be in the study for about two and a half years, and the study will involve visits to your study eye doctor's office about every 6 months. Your child will be asked to use eye drops every night for two years.
- The most likely risks to your child, which are expected to occur only rarely, are: blurry vision, skin irritation around the eyes, redness of the eyes or skin, stinging eyes, light sensitivity, an allergic reaction, dry skin and mouth, fast heartbeat, fever, and irritability.
- The possible benefits for your child are unknown, but that is what the study is trying to find out. Children who take part in this research study will add to new knowledge that may help other children with the same problem in the future.
- If you do not want your child to participate, there are other treatment options available for your child. Talk to your study eye doctor about: no treatment, regular eyeglasses or contact lenses, multi-focal contact lenses, rigid-gas permeable lenses at night, or bifocal glasses.





# LEGALLY AUTHORIZED REPRESENTATIVE (LAR)

Where we say "you" in this form, we mean a natural or adoptive parent, a legal custodian, or a legal guardian (collectively known as a "Legally Authorized Representative" or "LAR" for short). Where we say "your child" in this form, we mean the child under your direct care as the LAR.

#### WHAT IS INFORMED CONSENT?

We are asking you to allow your child to take part in this <u>research</u> study because your child has myopia (also known as nearsightedness). The goal of this research study is to learn things that may help children with myopia. Research is not the same as treatment. We want to find out what works best for treating your child and other children with this condition.

Your child's study doctor and nurse will be talking with you about this study and this form. You can take as much time as you need to think about whether or not you want your child to be in this study. You can also take a copy of this form with you to review with your child, your friends, family, or other doctors to help you decide. Please read this document carefully. Do not allow your child to be in this study unless all of your questions and your child's questions have been answered.

You do not have to allow your child to be in this study. If you decide that you do not want your child to be in this study, you and your child will not be treated differently. Also, you and your child's regular care will not be impacted.

#### WHO IS DOING THE STUDY?

Your child's eye doctor(s) will carry out this study. Their names are listed on the cover page of this form. The study is being done by the Pediatric Eye Disease Investigator Group. Your child's eye doctor is a member of this group. Funding for the study is being paid for by the National Eye Institute, which is part of the federal government. This funding will be used by the Jaeb Center for Health Research to organize the study and to pay your child's eye doctor for their work on the study. If one of the study doctors gets money or benefits from a company that makes the study drug (atropine) in this study, then they have to tell the Jaeb Center. The Jaeb Center has a policy to make sure that study doctors cannot work on this study if they get money or benefits that would influence how they do the study.

#### WHY IS THIS STUDY BEING DONE?

Nearsightedness means that vision is blurry when looking at far-away objects without glasses. This condition is also called myopia. Nearsightedness in a child is usually caused by an eye that is too long. If the eye continues to grow, children get more nearsighted. Once a child becomes nearsighted, it tends to get worse during childhood and teenage years, and stronger glasses are usually needed to correct the vision.





Some studies have shown that the low-dose atropine study eye drops may slow the progression of nearsightedness. The U.S. Food and Drug Administration (FDA) has not approved atropine for treating myopia (nearsightedness). Therefore, it is considered an experimental drug when used to treat myopia. The purpose of this study is to see if low-dose atropine eye drops can help prevent myopia from getting worse. The study will also see if any benefit lasts after the eye drops are stopped.

We expect about 400 children will take part in this study at about 10 different medical locations in the US.

#### WHO CAN PARTICIPATE IN THIS STUDY?

To take part in this study, your child must:

- be at least 5 years old, but younger than 13 years old
- have nearsightedness (myopia)
- have never had atropine eye drops to treat myopia before
- have never worn bifocals before
- have never worn special types of contact lenses used to slow myopia development
- have no known allergy to atropine

There are some other criteria your child must meet to be part of the study. Your study doctor will check if your child meets these or not. If your child meets the criteria but their current glasses do not meet the requirements for the study, the study will pay for new glasses or a change in your child's glasses, if you get them at the study doctor's office, LensCrafters or another study contracted optician.

Your child will be in the study for about 2 ½ years. You should NOT have your child be in the study if you are planning to move out of this area in the next 2 ½ years.

If your child is female, you should not have her take part in the study if she is pregnant or intending to become pregnant in the next 2 ½ years, or is nursing an infant. We will perform a pregnancy test at the time of enrollment if she has had a menstrual period. We will also perform pregnancy tests at follow up visits while your child is being treated with study medication (i.e. at (6-, 12-, 18- and 24-month visits), if she has had a menstrual period by then. We are required to do this testing even if you think there is no possibility that she is pregnant or could get pregnant during the study.

#### WHAT WILL HAPPEN IN THIS STUDY?

At the start of the study, all children will get placebo eye drops (without the atropine drug), also called artificial tears. These placebo eye drops contain no medication. They have no physical effect on the patient other than moistening the eye. Children will receive these drops in each eye every night for 2 to 4 weeks. Parents can put in the eye drops if the child is not able to. A smartphone app may be offered to parents to remind them to give the drops to their child every





night. Parents will need to record whether their child gets the eye drop every night. Children will need to return to their study eye doctor for another exam after using the eye drops for 2 to 4 weeks.

If your child has done well using these eye drops and still meets the criteria, a computer program will be used to select whether your child will be given study atropine eye drops or the placebo eye drops. This is like flipping a coin to decide which study group your child will be in, and is called randomization. Two out of three children will be given atropine eye drops. One out of three children will use placebo eye drops, which have no medicine. Neither you nor your doctor will know which group your child is in until the end of the study.

# Study Atropine 0.01% Eye Drops

Children in the study atropine eye drops group will receive one drop of low-dose atropine in each eye every night for 2 years. Your child will stop having the eye drops after 2 years. Your child will have a visit with the study doctor six months after stopping the drop. Your child will continue to wear glasses or contact lenses throughout the study.

# Placebo Eye Drops

Children in the placebo eye drops group will get one drop of placebo (artificial tears with no active drug) in each eye every night for 2 years. Your child will stop having the eye drops after 2 years. Your child will have a visit with the study doctor six months after stopping the drop. Your child will continue to wear glasses or contact lenses until throughout the study.

In both groups, your child will receive a new pair of glasses at 12 and 24 months and, if necessary, a lens change at 6 months and 18 months. The new glasses and lens changes will be provided at no cost to you if you get them at the study doctor's office, LensCrafters or another study contracted optician. The study will not pay for contact lenses or changes in contact lenses.

#### Visit Schedule

After starting in a study group, all children in the study will have visits with their study eye doctor at:

- 6 months
- 12 months
- 18 months
- 24 months
- 30 months

In addition, parents will get a phone call from their study eye doctor's office at:

- 2 weeks
- 3 months
- 9 months
- 15 months
- 21 months
- 27 months





The phone calls are to see if your child is experiencing any issues with treatment or to see if you have any questions about your child's participation in the study.

In the following table, you will find what will happen at each visit.

| Test | Enrollment | Randomization | 6 | 12 | 18 | 24 | 30 |
|---|---|---|---|---|---|---|---|
| Test | | 2-4 weeks | mos | mos | mos | mos | mos |
| Medical history | X | X | X | X | X | X | X |
| Pregnancy Test (for females | | | | | | | |
| who have had a menstrual | X | | X | X | X | X | |
| period) | | | | | | | |
| Questionnaire to evaluate the | | | | | | | |
| effect of eye drops on your | | X | X | X | X | X | |
| child | | | | | | | |
| Distance visual acuity to | | | | | | | |
| measure how well your child | | X | | | | | X |
| sees far away | | | | | | | |
| Near visual acuity to measure | | X | X | | | | |
| how well your child sees at near | | 71 | 1 | | | | |
| Accommodation (this tests the | | | | | | | |
| strength of your child's | | X | X | X | X | X | X |
| focusing system) | | | | | | | |
| Refraction (your doctor will | | | | | | | |
| manually measure your child's | X | | X | X | X | X | X** |
| eyeglasses prescription) | | | | | | | |
| Autorefraction (an automatic | | | | | | | |
| way to check your child's | | | | | | | |
| eyeglasses prescription; this | X | X* | X | X | X | X | X |
| will be done with dilating drops | | | | | | | |
| in the eyes) | | | | | | | |
| Biometry (to take | | _ | | | | | |
| measurements of your child's | X | X* | X | X | X | X | X |
| eyes) | | | | | | | |
| Prescribe artificial tears | X | | | | | | |
| Prescribe/refill study eye drops | | X | X | X | X | | |
| Stop study eye drops | | | | | | X | |
| Prescribe glasses or change in | X*** | | X*** | X | X*** | X | |
| spectacle lenses | 1 '1 1 | 1 1 .1 | | 1 6 | 11 | | |

<sup>\*</sup>Repeated at randomization if you child comes back more than 4 weeks from enrollment.

If you decide not to let your child take part in this study and do not sign this document, your child can continue receiving medical care not related to this study. If you decide to let your child

<sup>\*\*</sup>Standard refraction is not needed at 30 months if your child's vision has not changed much.

<sup>\*\*\*</sup> New glasses or a change in glasses will be provided at enrollment if needed. New glasses will be provided at 12 and 24 months. If needed, lenses will be changed at 6 and 18 months. The study will not pay for new or a change in contact lenses.





participate in the study, you can decide to stop your child's participation at any time. No penalty or loss of medical care will result from your decision not to let your child take part in this study.

#### WHAT ARE THE RISKS OF THIS STUDY?

If you decide to let your child take part in the study, your child will be at risk for the side effects listed below. Risks related to your child's normal medical care are not listed in this form. We encourage you to discuss these with your child's study doctor, your child's pediatrician, or another health care professional.

It is always possible that anyone taking a drug for the first time may have an allergic reaction. Also, there may be additional risks from the drug or the study procedures that are not known. If we find out that there are any new risks for your child, you will be told about them. You will be able to decide if you want your child to continue in the study based on this new information.

## **Eve Examinations:**

The risks and discomforts for the examinations will be the same whether or not your child is taking part in the study.

# **Study Drug(s):**

Studies have shown that the risks of using study atropine in both eyes for a long time depend on the atropine dose. This study is using a low dose of atropine (0.01%). This low dose of atropine has been used in other studies with very few side effects.

Study atropine (0.01%) may cause the following side effects, but these are rare:

- Blurry vision usually goes away after stopping the drops
- Skin irritation around the eyes
- Redness of the eyes or skin
- Stinging eyes
- Some light sensitivity children are encouraged to wear a hat with a brim and sunglasses
- Allergic reaction
- Dry skin and mouth
- Fast heart beat
- Fever

There are no known risks from taking placebo eye drops.

# **Risks to Confidentiality:**

This study will be capturing some information about your child that includes identifiable, personal information, like your child's date of birth. The study has procedures in place to protect that information. There is a chance that a loss of that protection could occur. This would be a loss of confidentiality. Please see the "How will my child's information be protected and kept confidential" section below for more information.



#### **Risks for Women:**

The risks of the drug used in this study on an unborn baby or a breastfeeding infant are unknown. For this reason, if your child is female, she cannot take part in the study if she is pregnant, planning to become pregnant within the next 2½ years, or nursing an infant. The study doctor will perform pregnancy tests before the study starts and at follow up visits during the two-year treatment period, if your child has had a menstrual period. The study doctors are required to do this even if you think there is no possibility that your child is pregnant or could get pregnant during the study. If the results of your child's pregnancy test are positive, they will only be told to you if your child gives permission. If your child becomes pregnant during the study, your child will stop taking the study drug but would be asked to stay in the study. If you are not comfortable with any of the following, then you should not allow your child to participate:

- your child having pregnancy tests
- the study doctor informing your child about positive pregnancy test results
- how the study doctor must get your child's permission to tell you pregnancy test results

#### **Washout Period:**

This study will involve a washout period without any eye drop treatment. The washout period will last 6 months. The risks associated with the washout period include potential increase in myopia or blurry distance vision without glasses. The washout period will help us understand if improvement in myopia is maintained after eye drops are discontinued.

# **Eye Drop Questionnaire**

At most follow-up visits, your child will be asked to complete a questionnaire assessing symptoms and the effect of eye drops on his or her health-related quality of life. If any questions make you or your child uncomfortable, then you or your child can refuse to answer.

# WHAT ARE THE BENEFITS OF MY CHILD TAKING PART IN THIS STUDY?

There may be a possible benefit to your child if you decide to let your child take part in the study, but that is what the study is trying to find out. Your child may receive no direct benefit from being in the study. Children who take part in this research study will add to new knowledge that may help other children with the same problem in the future.

#### ARE THERE OTHER OPTIONS THAN BEING IN THIS STUDY?

If you do not want your child to take part in this study, other options for your child include:

- No treatment
- Regular glasses or contact lenses
- Multi-focal contact lenses
- Rigid-gas permeable lenses at night
- Bifocal glasses

We encourage you to discuss these choices with your child's study doctor, your child's pediatrician, or another health care professional who has knowledge of myopia.



#### CAN MY CHILD STOP BEING IN THE STUDY?

You or your child can stop participation in this study at any time. If you or your child decide to stop being in this study, you and your child will not be treated differently. Also, you and your child's regular care will not be impacted. Please talk to your child's study doctor or staff so they know why you and your child are stopping the study and can help your child do so safely.

If we find out that there are any new risks, you will be told about them. You will be able to decide if you want your child to continue in the study based on this new information. The study may stop or the study doctor may decide to take your child out of the study at any time. You do not have to give permission for the study to stop or for the study doctor to remove your child from the study. You and your child will be told if this happens.

Some reasons why your child may be removed from the study include:

- The doctors feel that it is in the best interest of your child
- The doctors think that being in the study may cause your child harm
- If your child experiences an injury related to the study
- If your child needs additional or different medication
- If your child does not follow the study instructions

If your child is removed from the study or the study is stopped, your child may continue to receive care like your child normally would if your child were not in this study.

#### ARE THERE COSTS RELATED TO MY CHILD TAKING PART IN THE STUDY?

The costs of routine treatment, office visits, and tests that are part of your child's regular care will be billed to you or your child's insurance company like they normally would if your child were not in a study. The study will pay for the visits, procedures and drugs listed below. Any additional tests and procedures for standard care will be billed to you or your child's insurance company like they normally would. The study will pay for:

- Office visits that are part of the study (randomization visit, and visits at 6, 12, 18, 24, and 30 months).
- All eye drops used during the study (e.g. placebo artificial tears and atropine). At the end of the study, or if you decide to remove your child from the study, you must return any remaining eye drops to your child's eye doctor.
- Eyeglasses at enrollment (if needed), 12 months, and 24 months if you get them at the study doctor's office, LensCrafters or another study contracted optician. The study will also pay for lens changes at 6 and 18 months if the study requires it and the lenses come from the study doctor's office, LensCrafters or another study contracted optician. If your child has problems with schoolwork or reading, your child's eye doctor may prescribe bifocals. The study will pay for these bifocals if needed.





The study will not pay for:

- Eyeglasses obtained from somewhere other than the study doctor's office, LensCrafters or another study contracted optician.
- Contact lenses or a change in contact lenses.

#### IS THERE PAYMENT FOR TAKING PART IN THIS STUDY?

If you allow your child take part in the study, you will receive up to \$350 for participation. These payments will be paid as follows: \$50 to cover travel expenses for completion of the enrollment exam, randomization exam, and each study visit at 6, 12, 18, 24, and 30 months. These payments will be made by check or money card. If you have travel expenses that make it difficult for you to return for study visits, reimbursement may also be available for additional mileage at the Standard Mileage Rates specified by the government (for example, 54 cents per mile).

If you withdraw your child from the study, or if your child withdraws, you will still be paid for the visits that your child has completed. You will not receive extra payments for visits that are required as part of your child's normal care or for visits that are for treating an illness or injury.

# WHAT HAPPENS IF MY CHILD HAS AN ILLNESS OR INJURY FROM BEING IN THE STUDY?

If your child has an illness or injury that is related to your child's participation in the study, then you can get care for your child like you normally would. If your child has an emergency, please seek emergency care as soon as possible. Please tell the emergency doctor that your child is in a research study. Please also tell the study doctor about the emergency as soon as you can. The study will not provide costs for care or other expenses relating to illnesses or injuries. The costs of care for illnesses or injuries will be billed to you or your child's insurance company like they normally would. Your child's study doctor, the doctor's office, and the Jaeb Center are not offering payment for lost wages, direct losses, or indirect losses.

# CONTACT INFORMATION FOR QUESTIONS OR PROBLEMS

For questions about this study, a research illness or injury; or have concerns, suggestions or questions about the study, then contact the study doctor using the contact information on the first page of this form. You may also contact Pediatric Eye Disease Investigator Group (PEDIG) staff at 1-888-797-3344.

Contact the Jaeb Center for Health Research Institutional Review Board (IRB) Office at 813-975-8690 or <a href="mailto:irb@jaeb.org">irb@jaeb.org</a> if you:

- Have questions about your rights as a research participant
- Wish to talk about your concerns or suggestions about the research
- Want additional information about the research, or
- Want to provide comments about the research.





# HOW WILL MY CHILD'S INFORMATION BE PROTECTED AND KEPT CONFIDENTIAL?

As required by law, study related records with identifying information will be kept confidential. Safety measures for the access, security, and privacy of your child's information have been put in place by law. Unless the law requires it, your child's name, address, social security number, telephone number, or any other direct identifying information will not be used to identify your child.

# **Certificate of Confidentiality**

The National Institute of Health (NIH) has given us a Certificate of Confidentiality for this study. This adds special protection for study information that identifies your child and allows us, in some cases, to refuse to give out information that could identify your child without your consent. This could be done when the information is requested by a federal, state, local court or public agency. If your child needs medical help, we may still share your child's identifiable information. As described in this form or in other cases, we may share identifiable information. For example, if the government inspects us, they may see your child's identifiable information. Your child's study doctor and research team will follow local laws and will tell the local or state authorities:

- if certain diseases are present;
- if they suspect neglect, abandonment, or abuse of your child; and
- if your child's study doctor or research team learns that your child plans to harm self or others

#### **Purpose of Authorization**

We have rules to protect information about your child. Federal and state laws also protect your child's information. By signing this form you are giving your permission, called your "authorization," for the use and sharing of information protected by the law.

You must sign the <u>Protected Health Information Authorization</u> at the end of this form if you want your child to be in the study. When you sign the form, you give permission for the use and sharing of your child's Protected Health Information (PHI) for the study. PHI is health information that identifies your child. Your authorization is beneficial and important for the study. Without your authorization, your child will not be able to be in this study.

#### Using and Sharing Your Child's PHI

Your child's study doctor will collect information about your child. This information includes things learned from study procedures as well as your child's name, address, date of birth, and information from your child's medical records. These are examples of identifiable information. A code number will replace your child's name, address, telephone number, or social security number in the results given to the Jaeb Center for Health Research in Tampa, Florida.





The study doctor's office will <u>not</u> share study results that can identify your child except as explained in this form or when required by law. The Jaeb Center and your child's study doctor's office will guard the privacy of your child's study PHI.

Study results without the identifiable information may be shared in medical journals and at scientific meetings. Your child's records will be confidential. No one will share your child's identity in a medical journal or at a scientific meeting.

Results from the study will be sent to you in a newsletter upon completion of the research.

# Who Can Receive and Use Your Child's Study Information?

It is possible that people outside of this doctor's office and the Jaeb Center may need to see or receive your child's information from this study. Some examples include government agencies (such as the Food and Drug Administration), committees that monitor safety, other sites in the study, and companies that sponsor the study. In most cases the information <u>will</u> have a code number with it instead of your child's name, address, telephone number, or social security number.

There are some situations where the information will not have a code number but may include your child's name, address, telephone number, or social security number (PHI). If so, people outside this doctor's office who assist in your child's care may see your child's study PHI. They may not be covered by the law. Everyone who needs to see your child's information will be told it is confidential, but we cannot guarantee full confidentiality once it leaves the doctor's office.

#### **Other Considerations**

The information collected in the study may be used in future studies without additional permission from you. This may include research done by other researchers. The information that may be shared will <u>not</u> contain any information that could identify your child. There may still be a chance that someone could identify your child, but this is not likely. The study results will also be made public. These results will not have any information that could identify your child.

#### **Contact from the Jaeb Center**

Separately from your child's research data, the Jaeb Center for Health Research in Tampa, Florida will be provided with information on how to contact you.

- If your doctor's office is not able to locate you when they try to schedule your child's follow-up visit, the Jaeb Center may try to contact you through the alternative contact information you have given us. If this is not successful, the Jaeb Center may use the information you have given us to try to locate you through the use of a third-party search service.
- You may also receive updates about the study in the mail.

# **Study Eyeglasses**

Your child will receive eyeglasses as part of the study. They will be provided at no cost to you if you get them at the study doctor's office, LensCrafters or another study contracted optician.





Your child's study eye doctor may send you to LensCrafters or another contracted optician to get the new eyeglasses. In order to provide your child with new eyeglasses, the optician or LensCrafters will receive information on your child. Your child's name, birth date, and study identification number will be given to the optician who is making the eyeglasses. If your child is to receive study-paid eyeglasses through LensCrafters, this information will be given to LensCrafters by the Jaeb Center, via the EyeMed/Eye Care Plan of America website, to help process the making of your child's eyeglasses.

# **Clinical Trial Reporting**

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by law. This website will not include information that can identify your child. At most, the website will include a summary of the results. You can search this website at any time.

# **Can You Cancel Your Authorization?**

You may cancel your permission for the use and sharing of your child's study PHI at any time. You will need to contact your child's study doctors and give them a written notice of cancellation. When you cancel your permission or when you withdraw your child from the study directly, your child will no longer be a part of the study. No new information about your child will be gathered for the study except when there is a safety concern related to the study. If there is a safety concern, your child's entire medical record may need to be reviewed.

The Jaeb Center will receive all the information that was collected for the study up to the time that you cancel or withdraw your child from the study. The Jaeb Center will receive any new information about any safety concerns that may be related to the study.

# When Will the Use and Sharing of Your Child's PHI Stop?

Some of your child's study PHI does <u>not</u> have a code number with it. Your permission for the use and sharing of your child's PHI lasts 50 years from the date that you sign this form or until the end of the study, whichever comes first.

The rest of your child's study information does have a code number with it. When it is collected, it becomes part of a research report. Your permission for the use and sharing of this coded information will never end. This coded data <u>does not</u> have your child's name, address, telephone number, or social security number.

Some of your child's information from this study may be stored separately from or added to your child's medical record. You will not be able to see this information until the study ends. If your child's regular doctors require it for your child's care, they will be able to view it.





| Child's Full Name (printed): | |
|---|---|
| Legally Authorized Representatives (LARs) Pe | rmission |
| I, | _ (print name of legally authorized representative adividuals authorized to provide consent for the LARs (checkbox): |
| <ul> <li>□ Natural or Adoptive Parent</li> <li>□ Legal Custodian, or</li> <li>□ Legal Guardian</li> </ul> | |
| <ul> <li>you have read this informed consent form</li> <li>you have been given the chance to discuss th</li> <li>you authorize the use and sharing of your chast part of the study</li> </ul> | take part in this study. Your signature means that: the study and to ask questions to your satisfaction ild's protected health information that is collected icipate, you and your child can withdraw your y of this consent form |
| LAR Signature | Date |
| Investigator's Certification | |
| I certify that the LAR(s) named above are in child. I also certify that to the best of my know the nature, demands, risks, and benefits invol | |
| Investigator's Printed Name Investigator | r's Signature Date |